CLINICAL TRIAL: NCT04201002
Title: Squamous Cell Carcinoma Over Pilonidal Disease. A New Therapeutic Approach.
Brief Title: Surgery Plus Intraoperative Radiotherapy as Treatment for Squamous Cell Carcinoma Over Pilonidal Disease.
Status: Completed | Type: Observational
Sponsor: Hospital Provincial de Castellon (Other)
Responsible Party: Principal Investigator, Araceli Mayol Oltra, General Surgeon, Hospital Provincial de Castellon
Other Study IDs: HPCastellon
Record Dates: First submitted 2019-12-13; First posted 2019-12-16 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Squamous Cell Carcinoma; Pilonidal; Cyst, Malignant; Surgery
Keywords: Pilonidal sinus; Squamous cell carcinoma; Surgery; Intraoperative radiotherapy; Chemotherapy
MeSH Terms: conditions — Carcinoma, Squamous Cell; Cysts; Pilonidal Sinus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Resection plus intraoperative radiotherapy — En-bloc resection plus intraoperative radiotherapy

SUMMARY:
Background: Pilonidal sinus is a very common disease. Malignant transformation occurs in 0,1% of patients. The investigators present a case of squamous cell carcinoma arised from recurrent pilonidal disease, managed by multimodal treatment.

Case presentation: The investigators present a 70-year-old man with chronic pilonidal sinus. Inflammation had worsened in previous months and exploration revealed a large ulcerative mass which biopsy showed a squamous cell carcinoma. CT scan and MRI imaging showed tumoral invasion of the coccyx and both gluteus major muscles. Neoadjuvant radiotherapy, chemotherapy as radiosensitizer and surgery with intraoperative radiotherapy was decided in the multidisciplinary tumor committee. Post neoadjuvant therapy MRI showed partial response with a decrease of the mass but persistence of the coccyx infiltration.

Surgery consisted in en-bloc resection of the tumor with presacral tissues, coccyx and partial gluteal resection. Intraoperative radiotherapy was administered over the sacrum and in the bed of the coccyx resection. One week later, reconstructive surgery was practiced using a latissimus dorsi free flap, advancement of gluteal flaps and skin graft. Histological examination showed no residual tumor. The patient is currently asymptomatic and he has a satisfactory quality of life.

Conclusions: Although squamous cell carcinoma is rare, it must be suspected in patients with recurrent pilonidal disease. Diagnosis is done by histological examination of biopsies. This type of tumors have a high local recurrence rate. The investigators propose a multimodal treatment that includes neoadjuvant radiotherapy and chemotherapy as radiosensitizer and surgery plus intraoperative radiotherapy with the aim to decrease local recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma over pilonidal disease

Exclusion Criteria:

* Distant Metastases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We describe the diagnosis, treatment and follow-up of a patient with squamous cell carcinoma over pilonidal disease. The aim of the article is present the intraoperative radiotherapy plus en bloc surgery as a treatment in this cases with high recurrence rate.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Decrease in recurrence rate | 1 year
  Squamous cell carcinoma has a high recurrence rate, with surgery plus intraoperative radiotherapy we think it could decrease that recurrence rate.

CONTACTS AND LOCATIONS:
Overall Officials: Araceli Mayol Oltra, Principal Investigator — Consultant
Locations (2):
- Spain (2):
  - Hospital Provincial Castellon, Castellon, Castellon
  - Hospital Provincial Castellon, Castellon

IPD SHARING:
Plan to Share IPD: No